CLINICAL TRIAL: NCT05172479
Title: Prognostic Accuracy of qSOFA Score, SIRS Criteria, and EWSs for In-hospital Mortality Among Adult Patients Presenting With Suspected Infection to the Emergency Department (PASSEM): Protocol for an International Multicentre Prospective External Validation Cohort Study
Brief Title: Prognostic Accuracy of qSOFA, SIRS, and EWSs for In-hospital Mortality in Emergency Department
Acronym: PASSEM
Status: Completed | Type: Observational
Sponsor: Aseer Central Hospital (Other Government)
Collaborators: Armed Force Hospital Southern Region-Khamis Mushayt (AFHSR-KM) (Unknown); King Khalid University (KKU) (Unknown)
Responsible Party: Principal Investigator, Abdullah M Algarni, Family medicine consultant, Aseer Central Hospital
Other Study IDs: ACH-2
Record Dates: First submitted 2021-12-03; First posted 2021-12-29 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; qSOFA; SIRS; EWS; NEWS; NEWS2; MEWS; Emergency department
MeSH Terms: conditions — Sepsis; Shock, Septic; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Positive qSOFA: Adult patients with suspected infection and a qSOFA score ≥ 2 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of qSOFA score
- Negative qSOFA: Adult patients with suspected infection and a qSOFA score < 2 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of qSOFA score
- Positive SIRS: Adult patients with suspected infection and a SIRS criteria ≥ 2 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of SIRS criteria
- Negative SIRS: Adult patients with suspected infection and a SIRS criteria < 2 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of SIRS criteria
- Positive NEWS: Adult patients with suspected infection and a NEWS ≥ 5 or red score (i.e., a score of 3 in any one parameter) at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of NEWS
- Negative NEWS: Adult patients with suspected infection and a NEWS < 5 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of NEWS
- Positive NEWS2: Adult patients with suspected infection and a NEWS2 ≥ 5 or red score (i.e., a score of 3 in any one parameter) at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of NEWS2
- Negative NEWS2: Adult patients with suspected infection and a NEWS2 < 5 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of NEWS2
- Positive MEWS: Adult patients with suspected infection and a MEWS ≥ 5 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of MEWS
- Negative MEWS: Adult patients with suspected infection and a MEWS < 5 at the triage in the ED who are planned for hospitalization
  Interventions: Diagnostic Test: Measurement of MEWS

INTERVENTIONS:
Diagnostic Test: Measurement of qSOFA score — At the patient's arrival to the ED triage, the nurse will enter the patient's vital signs data into electronic data capture (EDC) system that will calculate the patient's qSOFA score.
  Other Names: quick Sequential Organ Failure Assessment (qSOFA)
  Groups: Negative qSOFA; Positive qSOFA
Diagnostic Test: Measurement of SIRS criteria — At the patient's arrival to the ED triage, the nurse will enter the patient's vital signs data into electronic data capture (EDC) system that will calculate the patient's SIRS criteria.
  Other Names: Systemic inflammatory response syndrome (SIRS)
  Groups: Negative SIRS; Positive SIRS
Diagnostic Test: Measurement of NEWS — At the patient's arrival to the ED triage, the nurse will enter the patient's vital signs data into electronic data capture (EDC) system that will calculate the patient's NEWS.
  Other Names: National Early Warning Score (NEWS)
  Groups: Negative NEWS; Positive NEWS
Diagnostic Test: Measurement of NEWS2 — At the patient's arrival to the ED triage, the nurse will enter the patient's vital signs data into electronic data capture (EDC) system that will calculate the patient's NEWS2.
  Other Names: National Early Warning Score 2 (NEWS2)
  Groups: Negative NEWS2; Positive NEWS2
Diagnostic Test: Measurement of MEWS — At the patient's arrival to the ED triage, the nurse will enter the patient's vital signs data into electronic data capture (EDC) system that will calculate the patient's MEWS.
  Other Names: Modified Early Warning Score (MEWS)
  Groups: Negative MEWS; Positive MEWS

SUMMARY:
Early identification of a patient with infection who may develop sepsis is of utmost importance. Unfortunately, this remains elusive because no single clinical measure or test can reflect complex pathophysiological changes in patients with sepsis. However, multiple clinical and laboratory parameters indicate impending sepsis and organ dysfunction. Screening tools using these parameters can help identify the condition, such as SIRS, quick SOFA (qSOFA), National Early Warning Score (NEWS), or Modified Early Warning Score (MEWS). The 2016 SCCM/ESICM task force recommended using qSOFA, while the 2021 Surviving Sepsis Campaign strongly recommended against its use compared with SIRS, NEWS, or MEWS as a single screening tool for sepsis or septic shock. We hypothesised that qSOFA has greater prognostic accuracy than SIRS and EWS (NEWS/NEWS2/MEWS).

DETAILED DESCRIPTION:
Over the past decade, medical advances in sepsis continued to focus on sepsis as a prevalent condition that accounts for 10% of admissions to intensive care units (ICUs) and is associated with a 10-20% in-hospital mortality rate. Standardised protocols and physician awareness have significantly improved survival, but mortality rates remain between 20% and 36%, with ~270,000 deaths annually in the United States. However, of patients with sepsis, 80% are treated in an emergency department (ED), and the remainder develops sepsis during hospitalisation with other conditions. In 2016, the Society of Critical Care Medicine/European Society of Intensive Care Medicine (SCCM/ESICM) task force redefined sepsis based on organ dysfunction and mortality prediction. Sepsis now is defined as life-threatening organ dysfunction caused by dysregulated host response to infection. This definition emphasises the complexity of the disease that cannot be explained by infection or body response to it. Acute change in Sequential Organ Failure Assessment (SOFA) score ≥2 indicates sepsis-related organ dysfunction, a predictor of excess in-hospital mortality. Systemic Inflammatory Response Syndrome (SIRS) and "severe sepsis" terms were omitted from the most recent definition. SIRS has been criticised for its poor specificity, while "severe sepsis" may underestimate sepsis's seriousness. A subset of patients may develop septic shock with underlying profound organ dysfunction and excess mortality. Clinically, septic shock is defined as persistent hypotension requiring vasopressors to maintain mean arterial pressure (MAP) ≥ 65 mm Hg and serum lactate level ≥ 2 mmol/L (18 mg/dL) despite adequate volume resuscitation. Early identification of a patient with infection who may develop sepsis is of utmost importance. Unfortunately, this remains elusive because no single clinical measure or test can reflect complex pathophysiological changes in patients with sepsis. However, multiple clinical and laboratory parameters indicate impending sepsis and organ dysfunction. Screening tools using these parameters can help identify the condition, such as SIRS, quick SOFA (qSOFA), National Early Warning Score (NEWS), or Modified Early Warning Score (MEWS). The 2016 SCCM/ESICM task force recommended using qSOFA, while the 2021 Surviving Sepsis Campaign strongly recommended against its use compared with SIRS, NEWS, or MEWS as a single screening tool for sepsis or septic shock. We hypothesised that qSOFA has greater prognostic accuracy than SIRS and EWS (NEWS/NEWS2/MEWS).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥18 years),
2. Suspected infection (based on the opinion of the emergency physician),
3. Planned for hospitalization,
4. Willing to give oral informed consent (if required by recruiting center's IRB).

Exclusion Criteria:

1. Presentation to ED is not due to infection (e.g., autoimmune diseases, myocardial infarction, stroke, venous thromboembolism, trauma, intoxication … etc.),
2. Pregnancy,
3. Transferred from another hospitals,
4. Code status is "Do-Not-Resuscitate" (DNR)
5. Elective admission through ED
6. Initial diagnosis of infection in the ED was not confirmed after finishing of the recruitment and follow-up phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients (age ≥18 years) presenting to the ED with suspected infection who planned to be hospitalized and willing to give informed consent (if required by recruiting center IRB) are eligible. A presumptive diagnosis of infection will be judged based on the opinion of the emergency physician upon the initial patient presentation to the ED. We will exclude patients with evidence of other causes of presentation to the ED other than infection (e.g., autoimmune diseases, myocardial infarction, trauma, …etc.), pregnant ladies, those who transferred from other hospitals, those not planned for hospitalization, or those who admitted electively to the hospital through ED. We will also exclude patients whose initial diagnosis of infection in the ED was not confirmed after the recruitment and follow-up.
Sampling Method: Probability Sample
Enrollment: 3274 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days
  Mortality rate during hospitalization of patient

SECONDARY OUTCOMES:
Intensive care unit admission | 30 days
  Number of participants admitted to an intensive care unit
Length of stay in the intensive care unit | 30 days
  Stay in intensive care unit >72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah M Algarni, MBBS, Principal Investigator — Aseer Central Hospital (ACH)
Locations (20):
- Bahrain (2):
  - Bahrain Defence Force Hospital, Riffa, Southern Governorate
  - King Hamad University Hospital, Al Muharraq
- Amiri Hospital, Kuwait City, Kuwait
- Armed Forces Hospital Oman, Muscat, Oman
- Hamad Medical Corporation, Doha, Qatar
- Saudi Arabia (12):
  - Aseer Central Hospital (ACH), Abhā, Aseer Province
  - Armed Force Hospital Southern Region-Khamis Mushayt (AFHSR-KM), Khamis Mushait, Aseer Province
  - King Fahad Specialist Hospital, Dammam, Eastern Province
  - Johns Hopkins Aramco Healthcare, Dhahran, Eastern Province
  - Royal Commission Hospital in Jubail, Jubail, Eastern Province
  - King Abdulaziz University Hospital, Jeddah, Makkah Al Mukarramah Province
  - King Fahd Armed Forces Hospital, Jeddah, Makkah Al Mukarramah Province
  - North Medical Tower, Arar, Northern Borders Province
  - King Abdullah bin Abdulaziz University Hospital (KAAUH), Riyadh, Riyadh Region
  - King Fahad Medical City (KFMC), Riyadh, Riyadh Region
  - King Saud Medical City (KSMC), Riyadh, Riyadh Region
  - Sulaiman Al-Habib Hospital, Riyadh
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)
- United Arab Emirates (2):
  - Sheikh Shakhbout Medical City, Abu Dhabi
  - Rashid Hospital, Dubai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Algarni AM, Alfaifi MS, Al Bshabshe AA, Omair OM, Alsultan MA, Alzahrani HM, Alali HE, Alsabaani AA, Alqarni AM, Alghanem SA, Al Mufareh BS, Almemari AM, Sindi AA, Ozturan IU, Alhadhira AA, Shujaa AS, Alotaibi AH, Awladthani MM, Alsaad AA, Almarshed AA, AlQahtani AM, Harris TR, Alyahya BA, Assiri SA, Abuzeyad FH, Kazim SN, Al-Fares AA, Almazroua FY, Marzook NT, Basri AA, Elsafti AM, Alalshaikh AS, Ozturan CA, Alawad YI, AlOmari A, Alkhateeb MA, Farooq MM, AlMutairi LA, Alasfour MM, Al Haber MI, Umar UA, Bokhary NH, Alqahtani SF, Almutairi A, Alyahya HF, Alzahrani WS, Alsalmi F, Omair AM, Alasmari FM, Alfifi SY, Al-Nujimi MS, Foroutan F. Prognostic accuracy of qSOFA score, SIRS criteria, and EWSs for in-hospital mortality among adult patients presenting with suspected infection to the emergency department (PASSEM) Multicenter prospective external validation cohort study protocol. PLoS One. 2024 Jan 17;19(1):e0281208. doi: 10.1371/journal.pone.0281208. eCollection 2024. PMID 38232095
- See also: Protocol preprint — https://www.medrxiv.org/content/10.1101/2022.03.19.22272537v1